CLINICAL TRIAL: NCT04386174
Title: Brain Activity in People With Chronic Neuropathic Pain and Spinal Cord Injury
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-1057-19
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Neuropathic Pain; Spinal Cord Injury
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Participants will be shown information about brain activity while trying different thinking strategies to change their experience of pain. Both groups will be shown brain activity, but the source of the brain activity information will differ between the groups.
  Interventions: Other: Neurofeedback
- Group B (Other): Participants will be shown information about brain activity while trying different thinking strategies to change their experience of pain. Both groups will be shown brain activity, but the source of the brain activity information will differ between the groups.
  Interventions: Other: Neurofeedback

INTERVENTIONS:
Other: Neurofeedback — Information about activity in pain-related regions of the brain will be shown to participants to determine if receiving this information is helpful in learning different thinking strategies (such as shifting attention, imagery, mantra meditation, etc.) that may help people with SCI change their experience of neuropathic pain.

SUMMARY:
The purpose of this research study is to learn more about how patterns of brain activity change during different thinking tasks and how these changes relate to the intensity and unpleasantness of the neuropathic pain that people with SCI experience.

DETAILED DESCRIPTION:
Neuropathic pain is a kind of pain that is caused by a disruption of the nervous system. Neuropathic pain is common among people with spinal cord injury (SCI), is often severe, and can interfere significantly with daily life. Current treatments do not eliminate neuropathic pain for most individuals. Therefore, it is important to identify other strategies that enable people with SCI to exert more control over their pain.

The purpose of this research study is to examine patterns of brain activity in people with SCI while they perform different thinking tasks. This study will help researchers understand how patterns of brain activity change during these tasks and how these tasks affect pain severity and unpleasantness. The information we learn in this study will help us create new treatment options to help people with SCI to manage their chronic neuropathic pain.

The study will take place over 2 days, separated by 1-3 weeks or so, depending on scheduling of study activities. The study should take approximately 1 hour on the first day (for a telephone interview), and up to 7.5 hours on the second day (for a visit to Kessler for functional magnetic resonance imaging, or fMRI).

In this study, participants will be asked to respond to a series of questions relating to their physical health, mental health, and pain history. The researchers may also review their medical records if needed to determine if it is safe for them to have an MRI. Those who qualify will visit Kessler and will be introduced to different thinking strategies that can be used to try to change the activity in the brain in areas that relate to the experience of pain. Participants will undergo 3 separate fMRI sessions. During the first session, the researchers will locate a pain-related region of the brain from which to gather information about brain activity. In the second and third sessions, the researchers will use fMRI to measure the activity in a pain-related region of the brain while the participant tries out different thinking strategies. While participants practice use of these strategies, they will be shown information about brain activity and will be asked to use this information as they try to become better at using the strategies. The researchers will also ask participants whether the experience of their pain (severity and unpleasantness) changed while they practiced these strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Right-handed
* Complete or incomplete chronic (>1 year) SCI classified as having a neurological level of C4 or below
* Chronic (≥3 month history) at- or below-level neuropathic pain
* Neuropathic pain of moderate or greater intensity (average intensity over the last week of ≥4 on an 11-point Numeric Rating Scale (NRS), where 0 = "no pain" and 10 = "worst pain imaginable")
* Neuropathic pain that is constant (present 7 days/week, 24 hours/day)
* Using a stable pain treatment regimen (not actively in process of starting a new pain treatment or changing dosage of an existing treatment)
* Able to understand verbal and written English
* Able and willing to comply with the study protocol, including availability for scheduled study procedures

Exclusion Criteria:

* Current non-neuropathic pain of severe intensity (average intensity over the last week of ≥7 on an 11-point NRS, where 0 = "no pain" and 10 = "worst pain imaginable")
* SCI due to malignancy
* Cognitive impairment that could interfere with learning (Mini-Mental State Exam score of <24)
* Current sacral, coccyx, or heel pressure injury
* Claustrophobia or fear of confined spaces
* Presence of any non-MRI compatible material in the body such as pacemakers or other implanted electrical devices, brain stimulators, particular types of dental implants, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves, and internal hearing aids [cochlear implants]), permanent eyeliner, implanted delivery pumps, or shrapnel fragments
* If female, currently pregnant
* Required use of non-MRI-compatible orthoses or devices (braces, ventilators, etc.)
* Current or past history of work as a welder or metal worker (because of possible small metal fragments in the eye of which they may be unaware)
* Inability to tolerate a supine position
* History (via self-report) of significant, uncontrollable spasticity while lying in supine position
* Progressive conditions that impact physical or cognitive functioning (metastatic cancer, multiple sclerosis, Parkinson Disease, Alzheimer's disease, etc.)
* History of traumatic brain injury
* Diagnosis of a psychiatric disorder such as post-traumatic stress disorder, schizophrenia or bipolar disorder
* History of substance abuse in the past six months
* Lack of intact sensation in the anterior shoulder (where stimuli will be applied during study procedures)
* Any other condition that would, in the opinion of the investigators, pose increased risk to the subject or affect the quality of data collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Brain activity | Immediately post-training session (1 day)
  Change in brain activity, as measured by Blood Oxygen Level Dependent (BOLD) signal

SECONDARY OUTCOMES:
Pain Intensity | Immediately post-training session (1 day)
  Intensity of pain rated on a 0-10 Numeric Rating Scale ranging from 0 = no pain to 10 = worst pain imaginable
Pain Unpleasantness | Immediately post-training session (1 day)
  Degree to which pain is unpleasant, rated on a 0-10 Numeric Rating Scale where 0 = not unpleasant at all to 10 = extremely unpleasant
Exit Interview | Immediately post-training session (1 day)
  Participants will be asked questions in a semi-structured interview to learn about their experiences trying to use the information on brain activity to help them learn strategies to self-manage pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No